CLINICAL TRIAL: NCT02970604
Title: PPARGC1β And CNTN4 Genotype as a Pharmacogenetic Assay of Thrombosis and Bleeding Risks - a Cross-Over Controlled Trial of Aspirin in Individuals at Increased Cardiovascular Risk.
Brief Title: PPARGC1β and CNTN4 Genotype Aspirin Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: RCSIMCT20152017
Record Dates: First submitted 2016-11-18; First posted 2016-11-22 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspirin (Experimental): Non-enteric coated Aspirin 75mg once daily for 7 days
  Interventions: Drug: Aspirin
- No treatment (No Intervention): No treatment for 7 days

INTERVENTIONS:
Drug: Aspirin — Non enteric coated aspirin
  Arms: Aspirin

SUMMARY:
Heart attacks and strokes are common causes of death worldwide. These events occur in part, due to increased activity of platelets, which cause clotting (thrombosis) within heart and brain blood vessels.

Anti-platelet therapies (e.g. aspirin) reduce the likelihood of platelet thrombosis and therefore protect against heart attacks and strokes. However serious bleeding into the gut and brain occurs in a number of individuals prescribed aspirin. Currently, there is no reliable method for assessing the relative risks of thrombosis versus bleeding in individual patients prior to or during aspirin therapy.

We have recently discovered that individuals with a particular genetic make-up, those with genetic variants in two genes called PPARGC1β and CNTN4, demonstrate more active (sticky) platelets. We then found that these same individuals suffered a greater number of cardiovascular events. Interestingly, low dose aspirin suppressed the excessive platelet stickiness and protected against heart attacks and strokes in these patients.

In this project, we aim to confirm and extend the above findings. We hope that testing for PPARGC1β and CNTN4 genetic variants will allow us to identify which patients will benefit from low dose aspirin therapy - i.e. receive protection from heart attacks and strokes, but not suffer any bleeding complications.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be male or female outpatients.
* Age must be greater than 18 years.
* Subjects must be able and willing to give written informed consent, and to comply with the requirements of this study protocol.
* Subjects must be at intermediate to high cardiovascular risk as determined by a calculated 5 year CVD risk of 5% or greater (calculated using the 1991 Anderson Framingham risk equation with adjustments as defined by the New Zealand Guidelines Group recommendations)

Exclusion Criteria:

* Age less than 18 years.
* Previous MI, stroke, transient ischaemic attack (TIA) or known CAD.
* Subjects who have any other significant disease or disorder (including concurrent malignancy) which, in the opinion of the investigator, may either put the subject at risk by participation in the study, or may influence the result of the study.
* Known history of, or documented positive hepatitis B or C or HIV infection
* AST or ALT ≥ 3 x ULN.
* Creatinine clearance (CrCl) < 60 mL/min measured by 24-hour urine collection or estimated by the Cockcroft and Gault formula.
* Female subjects who are pregnant or breast-feeding or considering becoming pregnant during the study, or with childbearing potential without using a medically accepted method of contraception (see notes 1-5 below)
* Patients already taking aspirin.
* Patients already taking anti-platelet agents (clopidogrel, ticagrelor etc), non-steroidal anti inflammatory drugs (NSAIDs), or anticoagulants (heparin, warfarin, dabigatran, etc).
* Patients who have a known intolerance to aspirin.
* Patients who have a contra-indication to aspirin as detailed below:

  * Hypersensitivity to salicylic acid compounds or prostaglandin synthetase inhibitors (e.g. certain asthma patients who may suffer an attack or faint and certain patients who may suffer from bronchospasm, rhinitis and urticaria) and to any of the excipients.
  * Active, or history of recurrent peptic ulcer and/or gastric/intestinal haemorrhage, or other kinds of bleeding such as cerebrovascular haemorrhages.
  * Haemorrhagic diathesis; coagulation disorders such as haemophilia and thrombocytopenia.
  * Patients who are suffering from gout.
  * Severe hepatic impairment.
  * Severe renal impairment.
  * Patients taking methotrexate used at doses >15mg/week.
* History of peptic ulcer disease or upper gastrointestinal bleeding.
* Subjects who have a history of drug or alcohol use that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Participants unlikely to comply well with study treatments or with the scheduled visits.
* Scheduled for procedures requiring general anaesthesia during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Urinary Thromboxane B2/Creatinine Ratio | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Alice Stanton, MB PhD, Principal Investigator — Royal College of Surgeons in Ireland
Locations (1):
- Royal College of Surgeons in Ireland, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No